CLINICAL TRIAL: NCT03515226
Title: Remote Training in Evidence-based Practices for Clinicians Who Work With Migrant Workers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges in recruiting eligible participants
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Pat Arean, Professor, Department of Psychiatry & Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00004268; 1P50MH115837-01 (NIH)
Record Dates: First submitted 2018-03-15; First posted 2018-05-03 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Depression
Keywords: workforce development; intelligent tutoring systems
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Training (Active Comparator): 20 hours of didactic education and training in CBT principles, depression assessment and cultural competency and 25 hours in dyad role playing of CBT manualized treatment sessions with supervision.
  Interventions: Behavioral: Traditional Training
- ITS based training (Experimental): Traditional training plus the addition of an algorithmic based training computer program that trains clinicians in clinical micro-competencies.
  Interventions: Behavioral: ITS based training

INTERVENTIONS:
Behavioral: ITS based training — Training using computerized adaptive training in addition to role play
  Arms: ITS based training
Behavioral: Traditional Training — Training using didactics and role plays
  Arms: Traditional Training

SUMMARY:
This study will compare training as usual to automated training using an intelligent tutoring system in training bachelors (BA) level social workers in cognitive behavioral therapy (CBT). The purpose of the study is to determine if time and cost of training front line clinicians in evidence-based treatments can be shortened, and if this new training model can reduce the need for clinicians to seek advice from experts.

DETAILED DESCRIPTION:
The University of Washington (UW) School of Social Work, in partnership with Heritage University's School of Social Work in Yakima Valley recently partnered to develop a training program for bachelors (BA) level Social Workers to address limited clinician capacity in rural primary care settings. Currently the curriculum is a combination of didactic training in telephone based cognitive behavioral therapy (CBT; 20 hours), role play training (25 hours), and guided supervision. The scalability of these programs is limited, however, by expert time to conduct training activities, clinician time away from work to engage in training activities, and the fact that even when clinicians participate in training, there is no guarantee they will certify. Adaptive learning, an educational method that uses adaptive algorithms to may be a potential solution to these problems in capacity building. These programs can tailor the educational experience to the needs of the trainee, reduce time in training, improve competence in complex decision-making and standardize training. This study builds on the existing research base on clinical training, and adds to it by designing and testing an intelligent tutoring system (ITS) based on adaptive learning algorithms. Both CBT experts (Aisenberg) and past CBT trainees (Heritage University School of Social Work) will partner with experts in educational software development (Popovic) to create the ITS, which will be compared to training as usual on time to training, competence and skill drift. The investigators hypothesize that capacity building through improved learnability (target mechanism) will result in enhanced clinical ability to deliver CBT elements competently, and in a shorter time-period, and that greater competence will result in better quality of care.

ELIGIBILITY:
Inclusion Criteria:

* BA level social work student
* Bilingual Spanish Speaking

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Arean, Principal Investigator — UWMC Psychiatry; Brenna Renn, PhD, Study Director — UWMC Psychiatry
Locations (1):
- University of Washington Department of Psychiatry and Behavioral Sciences, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will be creating a register of study outcomes for all projects under the UW ALACRITY center that researchers and request permission to access.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data for this study will be made available in January of 2021
Access Criteria: Any interested party who wishes to use our data for research or educational purposes may contact Dr. Renn who will review the request and provide access to information requested.

REFERENCES:
- [Derived] Lyon AR, Munson SA, Renn BN, Atkins DC, Pullmann MD, Friedman E, Arean PA. Use of Human-Centered Design to Improve Implementation of Evidence-Based Psychotherapies in Low-Resource Communities: Protocol for Studies Applying a Framework to Assess Usability . JMIR Res Protoc. 2019 Oct 9;8(10):e14990. doi: 10.2196/14990. PMID 31599736

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Training: 25 hours of didactic and simulated case role play training in CBT principles, depression assessment and cultural competency.
  Traditional Training: Training using didactics and role plays
Period: Overall Study
Arm/Group | Traditional Training | ITS Based Training
Started | 10 | 15
Completed | 8 | 11
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Traditional Training: 24 hours of didactic and simulated case role play training in CBT principles, depression assessment and cultural competency.
  Traditional Training: Training using didactics and role plays
- Total: Total of all reporting groups
Arm/Group | Traditional Training | ITS Based Training | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.63 (9.61) | 24.09 (8.63) | 24.74 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 0 | 7 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 8 | 16
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention Measure (AIM) - Goal Setting
Description: This is a four item measure of intervention acceptability; where each item is rated on a 1-5 scale, with 1 = not at all appropriate and 5 = very appropriate. The total scale range is 4-20. Each group will be compared on the degree they find the specific clinical skill acceptable to use after they complete the training. We administered the AIM twice asking the students to respond to the acceptability of goal setting as a clinical skill and of identifying challenges as a clinical skill. This section reports on goal setting.
Time Frame: This measure will be administered to participants in each training group after they complete the 25 hours of training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Training | ITS Based Training
Number analyzed (Participants) | 8 | 11
score on a scale
  Pre-Training | 17.88 (0.99) | 17.64 (1.43)
  Post-Training | 17.63 (1.69) | 18.27 (2.61)

2. Primary Outcome: Acceptability of Intervention Measure (AIM) - Identifying Challenges
Description: This is a four item measure of intervention acceptability; where each item is rated on a 1-5 scale, with 1 = not at all appropriate and 5 = very appropriate. The total scale range is 4-20. Each group will be compared on the degree they find the specific clinical skill acceptable to use after they complete the training. We administered the AIM twice asking the students to respond to the acceptability of goal setting as a clinical skill and of identifying challenges as a clinical skill. This section reports on identifying challenges.
Time Frame: This measure will be administered to participants in each training group after they complete the 25 hours of training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Training | ITS Based Training
Number analyzed (Participants) | 8 | 11
score on a scale
  Pre-Training | 16.75 (1.39) | 17.73 (3.44)
  Post-Training | 16.25 (1.28) | 17.82 (1.72)

3. Primary Outcome: Intervention Appropriateness Measure (IAM) - Goal Setting
Description: This is a four item measure of intervention appropriateness; where each item is rated on a 1-5 scale, with 1 = not at all appropriate and 5 = very appropriate. The total range for this measure is 4-20. Each group will be compared on the degree they find the specific clinical skill appropriate to use after they complete the training. We administered the IAM twice asking the students to respond to the acceptability of goal setting as a clinical skill and of identifying challenges as a clinical skill. This section reports on goal setting.
Time Frame: This measure will be administered to participants in each training group after they complete the 25 hours of training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Training | ITS Based Training
Number analyzed (Participants) | 8 | 11
score on a scale
  Pre-Training | 18.25 (1.75) | 18.55 (1.63)
  Post-Training | 17.88 (2.23) | 18.82 (1.54)

4. Primary Outcome: Intervention Appropriateness Measure (IAM) - Identifying Challenges
Description: This is a four item measure of intervention appropriateness; where each item is rated on a 1-5 scale, with 1 = not at all appropriate and 5 = very appropriate. The total scale range is 4-20. Each group will be compared on the degree they find the specific clinical skill appropriate to use after they complete the training. We administered the IAM twice asking the students to respond to the acceptability of goal setting as a clinical skill and of identifying challenges as a clinical skill. This section reports on identifying challenges.
Time Frame: This measure will be administered to participants in each training group after they complete the 25 hours of training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Training | ITS Based Training
Number analyzed (Participants) | 8 | 11
score on a scale
  Pre-Training | 16.38 (1.19) | 18.82 (2.27)
  Post-Training | 17.13 (1.81) | 18.27 (1.90)

5. Primary Outcome: Feasibility of Intervention Measure (FIM) - Goal Setting
Description: This is a four item measure of intervention feasibility; where each item is rated on a 1-5 scale, with 1 = not at all appropriate and 5 = very appropriate. The total scale range is 4-20. Each group will be compared on the degree they find the specific clinical skill feasible to use after they complete the training they participated in. We administered the FIM twice asking the students to respond to the feasibility of goal setting as a clinical skill and of identifying challenges as a clinical skill. This section reports on goal setting.
Time Frame: This measure will be administered to participants in each training group after they complete the 25 hours of training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Training | ITS Based Training
Number analyzed (Participants) | 8 | 11
score on a scale
  Pre-Training | 16.88 (2.23) | 17.09 (2.17)
  Post-Training | 17.13 (1.46) | 18.91 (1.64)

6. Primary Outcome: Feasibility of Intervention Measure - Identifying Challenges
Description: This is a four item measure of intervention feasibility; where each item is rated on a 1-5 scale, with 1 = not at all appropriate and 5 = very appropriate. The total scale range is 4-20. Each group will be compared on the degree they find the specific clinical skill feasible to use after they complete the training they participated in. We administered the FIM twice asking the students to respond to the feasibility of goal setting as a clinical skill and of identifying challenges as a clinical skill. This section reports on identifying challenges.
Time Frame: This measure will be administered to participants in each training group after they complete the 25 hours of training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Training | ITS Based Training
Number analyzed (Participants) | 8 | 11
score on a scale
  Pre-Training | 15.88 (2.30) | 17.73 (2.45)
  Post-Training | 15.63 (1.69) | 18.27 (1.68)

7. Primary Outcome: Intervention Usability Scale (IUS) - Goal Setting
Description: The IUS is a 10-item measure with a possible total score ranging from 0 to 100; higher scores indicate a more usable intervention. Although this measure has not yet been normed as a measure of intervention usability, the System Usability Scale upon which the IUS is based defines scores of 70 or above as indicative of acceptable usability.
Time Frame: This measure will be administered to participants in each training group after they complete the 25 hours of training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Training | ITS Based Training
Number analyzed (Participants) | 8 | 11
score on a scale
  Pre-Training | 28.25 (3.85) | 28.27 (3.61)
  Post-Training | 30.13 (5.03) | 30.82 (4.02)

8. Primary Outcome: Intervention Usability Scale (IUS) - Identifying Challenges
Description: as for outcome 7
Time Frame: This measure will be administered to participants in each training group after they complete the 25 hours of training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Training | ITS Based Training
Number analyzed (Participants) | 8 | 11
score on a scale
  Pre-Training | 26.75 (4.30) | 27.91 (4.55)
  Post-Training | 28.88 (4.09) | 29.27 (5.10)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Traditional Training | ITS Based Training
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/8 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT03515226/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT03515226/ICF_001.pdf